CLINICAL TRIAL: NCT04012073
Title: Individualized Positive End-expiRatory Pressure Guided by End-Expiratory Lung Volume in Moderate-to-severe Acute resPiratory Distress Syndrome.The IPERPEEP Study
Brief Title: Individualized Positive End-expiratory Pressure Guided by End-expiratory Lung Volume in the Acute Respiratory Distress Syndrome
Acronym: IPERPEEP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely terminated following the funder's decision to withdraw financial support.
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: ClinicalTrialCenter (Unknown); FerrarioDati (Unknown); General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANT-IPE-18-006
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Positive end-expiratory pressure; Ventilator-induced lung injury; Mechanical ventilation; Respiratory mechanics
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury | interventions — Neuromuscular Blocking Agents; Prone Position; Airway Extubation

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified according to Recruitment/cmH2O ≥ or < 19 ml/cmH2O across the range between the lowest and highest PEEP tested during the initial PEEP trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IPERPEEP (Experimental): End expiratory lung volume (EELV) will be measured at each step during a 5-step decremental PEEP trial.
  PEEP will be ≥5 cmH2O and set to ensure the maximum recruitment observed in the PEEP trial, with a maximum permitted PPLAT of 30 cmH2O.
  In particular, when interpreting the results of the PEEP trial, recruitment-to-inflation (RI) ratio calculated across two adjacent PEEP levels will drive PEEP setting.
  * RI≥1.5 between two PEEP levels will lead to the setting of the higher PEEP.
  * RI<0.5 will lead to the setting of the lower PEEP value.
  * In case of RI≥0.5 and <1.5, the choice among two adjacent PEEP levels will be left to the attending physician, who will indicate the set PEEP in order to best balance between the commitment of limiting total, static and dynamic strain and of optimizing oxygenation and haemodynamics.
  Interventions: Device: Invasive Mechanical ventilation; Drug: Neuromuscular Blocking Agents; Procedure: Prone positioning; Procedure: Resume of spontaneous breathing; Procedure: Rescue treatments; Procedure: Weaning from PEEP; Procedure: Weaning from mechanical ventilation; Procedure: Extubation
- EXPRESS (Active Comparator): PEEP set so that the plateau pressure is within the following limits: 28 cmH2O≤Pplat≤ 30 cmH2O
  Interventions: Device: Invasive Mechanical ventilation; Drug: Neuromuscular Blocking Agents; Procedure: Prone positioning; Procedure: Resume of spontaneous breathing; Procedure: Rescue treatments; Procedure: Weaning from PEEP; Procedure: Weaning from mechanical ventilation; Procedure: Extubation

INTERVENTIONS:
Device: Invasive Mechanical ventilation — Volume-control ventilation with tidal volume will be set at 6 mL/Kg of predicted body weight, respiratory rate to maintain pH>7.30 and PaCO2<50 mmHg and FiO2 will be set to achieve a SpO2>88-95%.
  In case of hypercapnia with Ph<7.30 despite a respiratory rate=30-35, an increase in tidal volume up to 8 ml/kg will be allowed.
  In both groups, the assigned ventilation protocol will be followed for a minimum of 72 hours from randomization and any time fully controlled ventilation is deemed necessary by the attending physician up to 14 days from randomization. After 14 days from randomization, PEEP will be set according to the clinical practice of each institution.
  After 72 hours from the study protocol, the PEEP setting protocol according to the assigned treatment will be resumed at any time within 14 days from enrolment if fully controlled ventilation is established, according to the decision of the attending physician in charge.
Drug: Neuromuscular Blocking Agents — All patients will receive NMBA for 48 hours after the enrolment. The decision to stop NMBA administration after 48 hours will be left to the attending physician, but muscle paralysis will be strongly encouraged if PaO2/FiO2 ratio remains lower than 80-100 mmHg. NMBA administration will be resumed anytime deemed necessary by the attending physician.
Procedure: Prone positioning — Prone positioning will be used in all enrolled patients as a standard of care: the decision about the timing and the duration of prone position sessions will be left to the attending physician and the time spent by the patient in the prone and in the supine position will be recorded: PEEP will be re-set according to the protocol of the allocated treatment anytime patient's position is changed.
Procedure: Resume of spontaneous breathing — Assist/control and assist ventilation will be allowed after 72 hours from the enrolment if deemed appropriate by the attending physician.
  During spontaneous breathing, PEEP will be set according to the decision of the attending physician and the practice of each institution: however, in order to standardize the treatments, moderate PEEP (10-15 cmH2O) will be encouraged in case of moderate hypoxemia (PaO2/FiO2<150 mmHg) in control group, while PEEP close to the value set during controlled ventilation according to the treatment protocol but <15 cmH2O will be suggested in the intervention group.
  During assist/control and assisted ventilation, PEEP will never be higher than the last PEEP set according to the assigned protocol during controlled ventilation.
  Fully controlled mechanical ventilation will be resumed any time during the study period if the patient meets the criteria described above or any time deemed necessary by the physicians in charge
Procedure: Rescue treatments — Recruitment maneuvers, extracorporeal membrane oxygenation (ECMO), extracorporeal CO2 removal (ECCO2-R) after randomization will be allowed in both groups as rescue therapies and according to the decision of attending physicians: any of these procedures will be accurately recorded on the case report form.
Procedure: Weaning from PEEP — In order not to delay weaning from mechanical ventilation, when a patient is managed with assist/control or assist ventilation with PEEP higher than 8 cmH2O, a daily PEEP weaning trial will be performed whether PaO2/FIO2 ratio>150 mm Hg and FIO2<0.5: PEEP will be decreased to 8-5 cm H2O and arterial blood gas will be sampled after 20 -0 minutes. Previous ventilatory settings will be resumed if during the procedure transcutaneous oxyhemoglobin saturation decreases below 88%, PaO2/FIO2 falls below 150 mm Hg or if the patient experiences abnormal changes in respiratory rate or other clinical signs suggestive of respiratory distress.
  When PaO2/FIO2 is no lower than 200 mm Hg at PEEP≤8 cmH2O, the patient will be considered to have acceptable gas exchange on 8-5 cmH2O of PEEP and will be deemed capable to tolerate this setting
Procedure: Weaning from mechanical ventilation — A 30-120-minute spontaneous breathing trial will be initiated as the following criteria are met and whether the patient tolerates fully assist ventilation with PEEP≤8 cmH2O for at least 4 hours without experiencing hypoxemia (SpO2<88% or PaO2/FiO2<150mmHg):
  * improvement or resolution of the underlying cause of acute respiratory failure
  * normal sensorium
  * correction of arterial hypoxemia (PaO2 ≥ 60 mmHg at a FiO2 ≤ 0.4 with PEEP ≤ 8 cmH2O);
  * absence of fever (≥ 38 °C) or sepsis;
  * blood hemoglobin concentration of 7 g/dL or more;
  * hemodynamic stability
  For the purpose of the study, success of the spontaneous breathing trial will be defined as presence of the following criteria:
  * respiratory rate < 35/min,
  * arterial oxygen saturation ≥ 90%,
  * heart rate < 120/min,
  * systolic blood pressure > 90 and < 160 mmHg
  * adequate cough. If the spontaneous breathing trial is successful, the patient will be extubated.
Procedure: Extubation — Each extubated patient will undergo oxygen therapy via high flow nasal cannula (maximum flows tolerated and FiO2 titrated to obtain 96%>SpO2>92%). Pre-emptive noninvasive ventilation (NIV) after extubation will be allowed in prolonged to wean patients (i.e. more than 3 SBT failure or more than 7 days from the first spontaneous breathing trial to being extubated) if deemed necessary by the physician in charge.
  In case of respiratory failure during oxygen therapy via high flow nasal cannula after extubation and, a rescue NIV trial will be allowed before intubation in both groups at the discretion of the attending physician.

SUMMARY:
During the acute respiratory distress syndrome (ARDS), patients' response to positive end-expiratory pressure (PEEP) is variable according to different degrees of lung recruitability. The search for a tool to individualize PEEP on the basis of patients' individual response is warranted.

Measurement of end-expiratory lung volume (EELV) by the nitrogen washin-washout technique, bedside available from recent ICU ventilators, has been shown to reliably estimate PEEP-induced alveolar recruitment and may therefore help titrate PEEP on patient's individual requirements.

The authors designed an open-label, multicenter, randomized trial to test whether an individualized PEEP setting protocol driven by EELV may improve a composite clinical outcome in patients with moderate-to-severe ARDS.

DETAILED DESCRIPTION:
ARDS patients with a PaO2/FiO2 ratio equal or below 150 mmHg (during mechanical ventilation with PEEP 5 cmH2O) will be enrolled within 24 hours from endo-tracheal intubation.

To standardize lung volumes at study initiation, all patients will undergo mechanical ventilation with tidal volume set at 6 ml/kg of predicted body weight and PEEP set to obtain a plateau pressure within 28 and 30 cmH2O for thirty minutes (Express PEEP).

Afterwards, a 5-step decremental PEEP trial will be conducted (Express PEEP to PEEP 5 cmH2O), and EELV will be measured at each step. PEEP-induced alveolar recruitment will be calculated for each PEEP range as the difference between PEEP-induced change EELV and the predicted increase in lung volume due to PEEP (PEEP-induced overdistension, equal to the product of respiratory system compliance and PEEP change).

Patients will be then randomized to receive mechanical ventilation with PEEP set according to the optimal recruitment observed in the PEEP trial (IPERPEEP arm) trial or according to the Express strategy (Control arm, PEEP set to achieve a plateau pressure of 28-30 cmH2O).

In both groups, tidal volume size, the use of prone positioning and neuromuscular blocking agents will be standardized.

Primary endpoint of the study is a composite clinical outcome incorporating in-ICU mortality, 60-day ventilator free days and the area under the curve of serum Interleukin 6 over the course of the initial 72 hours.

Primary and secondary endpoints will also be analyzed in subgroups, as defined below:

* ∆EELV5-16/FRC ≥ 73% [18] during the PEEP trial
* ∆EELV5-16/FRC < 73%[23] during the PEEP trial
* Recruitment-to-inflation ratio (RI) ≥ 1 and <1 across the range between the lowest and highest PEEP tested during the PEEP trial
* P/F ratio<100 mmHg at study inclusion
* IL-6>400 pg/ml at study inclusion

ELIGIBILITY:
Eligibility inclusion criteria, according to the ARDS Berlin definition, will be assessed within the first 24 hours from the initiation of invasive mechanical ventilation:

1. Acute respiratory failure within 1 week of a known clinical insult or new or worsening respiratory symptoms;
2. Bilateral infiltrates at the chest x-ray or CT scan, not fully explained by effusions, lobar/lung collapse, or nodules;
3. Respiratory failure not fully explained by cardiac failure or fluid overload; objective assessment required to exclude hydrostatic edema if no risk factor present.
4. PaO2/FiO2 ratio≤150 mmHg after 30 mins - 1 hour of mechanical ventilation with PEEP=5 cmH2O.
5. Written informed consent.

Exclusion Criteria:

1. Pregnancy;
2. Pneumothorax;
3. Acute brain injury;
4. Clinical signs of history of decompensated heart failure (New York Heart Association class 3-4 before the acute phase of the disease or documented ejection fraction<35% or pulmonary capillary wedge pressure>18 mmHg) or acute coronary syndrome;
5. Intubation as a result of an acute exacerbation of chronic pulmonary disease: chronic obstructive pulmonary disease, asthma, cystic fibrosis, etc;
6. Clinically evident intrinsic PEEP (≥2 cmH2O) during screening visit (End-expiratory pause to achieve Flow=0);
7. BMI>35;
8. BMI<15 or body weight<35 Kg;
9. Any chronic disease requiring long-term oxygen therapy or mechanical ventilation at home;
10. Neuromuscular disease of any kind;
11. Severe chronic liver disease (Child-Pugh C or worse);
12. Bone marrow transplantation or chemotherapy-induced neutropenia;
13. History of liver or lung transplant;
14. Decision to withhold life-sustaining treatment;
15. Need for therapy with inhaled nitric oxide due to documented pulmonary arterial hypertension;
16. Life-threatening hypoxemia deemed to require extracorporeal membrane oxygenation (ECMO);
17. Presence of documented barotrauma;
18. High risk of mortality within 3 months from other than ARDS (severe neurological damage, age >85 years and cancer patients in terminal stages of the disease).
19. Persistent hemodynamic instability, intractable shock (norepinephrine>1 mcg/kg/h and/or blood lactate>5 mmol/L and/or considered too hemodynamically unstable for enrolment in the study by the patient's managing physician).
20. More than 24 hours from endotracheal intubation to the time of the screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Composite clinical outcome that incorporates ICU mortality, 60-day ventilation-free days (VFD60) and the Area Under the Curve of the InterLeukin-6 serum concentration (IL6AUC) during the first 72 hours of observation | 60 days
  Composite clinical outcome that incorporates ICU mortality, 60-day ventilation-free days (VFD60) and the Area Under the Curve of the InterLeukin-6 serum blood cytokine concentration (IL6AUC) during the first 72 hours of observation. Every participant in the treatment group will be compared with every participant in the control group and assigned a score resulting from each comparison. Mortality takes precedence over VFD60, which takes precedence over IL6AUC. Two VFD60's will be considered different for the purpose of scoring only if their difference is larger than 5 days. Similarly, two IL6AUC's measurements will be considered different only if their difference exceeds 10% of the smaller of the two. These individual-comparison scores are added up to obtain the cumulative score primary endpoint for each participant. The sum of scores for patients in the treatment group is compared to the sum of scores of subjects in the control group and compared according by use of Mann-Whitney test

SECONDARY OUTCOMES:
In-ICU mortality | 90 days
  Mortality at ICU discharge
In-Hospital mortality | 90 days
  Mortality at hospital discharge
90-day mortality | 90 days
  Mortality at 90 days from randomization
28-day Ventilator free days | 28 days
  The days spent without ventilator assistance within 28 days from randomization
60-day Ventilator free days | 28 days
  The days spent without ventilator assistance within 60 days from randomization
Time to successful weaning | 90 days
  The time from enrolment to successful liberation from mechanical ventilation
Time spent on assisted ventilation after the enrolment | 28 days
  The time spent on assisted ventilation on 28-day basis
AUC IL-6 | 72 hours
  Area under the curve (AUC) of serum interleukin 6 in the initial 72 hours of treatment
AUC IL-8 | 72 hours
  Area under the curve (AUC) of serum interleukin 8 in the initial 72 hours of treatment
AUC TNF | 72 hours
  Area under the curve (AUC) of serum tumor necrosis factor in the initial 72 hours of treatment
Plateau pressure | 72 hours
  Plateau pressure during the assigned treatment
Total Lung stress-End-inspiratory transpulmonary pressure derived from elastance ratio | 72 hours
  Total increase in transpulmonary pressure due to tidal volume and PEEP during the assigned treatment
Static stress | 72 hours
  Total increase in transpulmonary pressure due to PEEP during the assigned treatment
Set PEEP | 72 hours
  Set PEEP during the assigned treatment
Set PEEP variability | 72 hours
  Ratio of standard deviation to mean PEEP during the assigned treatment
End-expiratory transpulmonary pressure | 72 hours
  Directly measured end-expiratory transpulmonary pressure during the assigned treatment
Dynamic stress-Transpulmonary driving pressure | 72 hours
  Total increase in transpulmonary pressure due to tidal volume during the assigned treatment
Respiratory system driving pressure | 72 hours
  The difference between Plateau Pressure and total PEEP during the assigned treatment
Respiratory system compliance | 72 hours
  Ratio of tidal volume to respiratory system driving pressure during the assigned treatment
Respiratory system compliance normalized to predicted body weight | 72 hours
  Ratio of respiratory system compliance and predicted body weight during the assigned treatment
Lung compliance | 72 hours
  Ratio of tidal volume to transpulmonary driving pressure during the assigned treatment
Dynamic strain | 30 minutes
  Ratio of tidal volume to end-expiratory aerated volume (end-expiratory lung volume plus PEEP-induced alveolar recruitment) at study start
Static strain | 30 minutes
  Ratio of PEEP-induced overdistension volume to end-expiratory aerated volume (end-expiratory lung volume plus PEEP-induced alveolar recruitment) at study start
Oxygenation | 72 hours
  Ratio of PaO2 to FiO2 during the assigned treatment
Oxygenation stretch index | 72 hours
  Ratio of PaO2/FiO2 to respiratory system driving pressure during the assigned treatment
Carbon dioxide | 72 hours
  Arterial pressure of CO2 during the assigned treatment
Heart rate | 72 hours
  Heart rate during the assigned treatment
Arterial pressure | 72 hours
  Mean arterial pressure during the assigned treatment
Simplified organ failure assessment | 28 days
  Simplified organ failure assessment (SOFA) after randomization
Catecholamine requirements per day | 72 hours
  Catecholamin administration ad dosage during the assigned treatment
Organ failure | 28 days
  Organ failure free days on a 28-day basis, as defined by the simplified organ failure assessment (SOFA)
Need for rescue recruitment maneuvers | 72 hours
  The proportion of patients needing rescue recruitment maneuvers during the assigned treatment
Nedd for rescue extra-corporeal membrane oxygenation | 90 days
  The proportion of patients needing rescue extra-corporeal membrane oxygenation due to persistent hypoxemia
Nedd for tracheostomy | 90 days
  The proportion of patients needing tracheostomy to enhance the weaning process

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Chair — Fondazione Policlinico Universitario A. Gemelli IRCCS; Università Cattolica del Sacro Cuore; Domenico Luca Grieco, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS; Università Cattolica del Sacro Cuore
Locations (10):
- Italy (10):
  - Policlinico di Bari, Bari
  - Policlinico Sant'Orsola, Bologna
  - Azienda ospedaliero-universitaria Mater Domini, Catanzaro
  - SS. Annunziata hospital, Chieti
  - Azienda ospedaliera universitaria di Ferrara-arcispedale Sant'Anna, Ferrara
  - Ospedale San Martino, Genova
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Gerardo, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available upon a reasonable request
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Grieco DL, Maggiore SM, Bellani G, Spadaro S, Spinelli E, Tonetti T, Menga LS, Pozzi M, Battaglini D, Di Mussi R, Bruni A, De Gaetano A, Iovino CG, Brioni M, Mojoli F, Foti G, Volta CA, Pelosi P, Navalesi P, Grasso S, Ranieri VM, Antonelli M; IPERPEEP study group. Individualized positive end-expiratory pressure guided by end-expiratory lung volume in early acute respiratory distress syndrome: study protocol for the multicenter, randomized IPERPEEP trial. Trials. 2022 Jan 20;23(1):63. doi: 10.1186/s13063-021-05993-0. PMID 35057852
- [Derived] Santa Cruz R, Villarejo F, Irrazabal C, Ciapponi A. High versus low positive end-expiratory pressure (PEEP) levels for mechanically ventilated adult patients with acute lung injury and acute respiratory distress syndrome. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD009098. doi: 10.1002/14651858.CD009098.pub3. PMID 33784416